CLINICAL TRIAL: NCT07164352
Title: Effect of Breathing Exercises on Pain, Dyspnea, and Functionality in Terminal-Stage Cancer Patients Receiving Palliative Care - Master's Thesis, İstanbul Atlas University, Graduate School, Dept. of Physical Medicine and Rehabilitation
Brief Title: Effect of Breathing Exercises on Pain, Dyspnea, and Function in Terminal-Stage Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Fatma Nur Yildiz, Physiotherapist, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS-FTR-FNY-01
Record Dates: First submitted 2025-05-23; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Palliative Patients; Terminal Malignant Tumors; Breathing Techniques
Keywords: Palliative Care; Terminal Stage Cancer; Breathing Exercises
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragmatic and pursed-lip breathing exercises supervised by a physiotherapist (Experimental): Participants in this arm receive supervised breathing exercises performed with a physiotherapist, focusing on diaphragmatic and pursed-lip breathing techniques.
  Interventions: Behavioral: Breathing Exercises
- Brochure Education Only (Active Comparator): Participants in this arm receive an informational brochure that explains breathing exercises, but no supervised exercise is provided.
  Interventions: Behavioral: Informational Brochure

INTERVENTIONS:
Behavioral: Breathing Exercises — Diaphragmatic and pursed-lip breathing exercises supervised by a physiotherapist.
  Arms: Diaphragmatic and pursed-lip breathing exercises supervised by a physiotherapist
Behavioral: Informational Brochure — A brochure providing education about breathing exercises for cancer patients.
  Arms: Brochure Education Only

SUMMARY:
This study aims to evaluate the effects of supervised breathing exercises on pain, dyspnea, and functionality in terminal-stage cancer patients receiving palliative care. Participants in the intervention group receive diaphragmatic and pursed-lip breathing exercises under the guidance of a physiotherapist, while the control group receives only an educational brochure. The study compares pre- and post-intervention outcomes between both groups.

DETAILED DESCRIPTION:
This randomized controlled trial aims to investigate the effects of diaphragmatic and pursed-lip breathing exercises on pain, dyspnea, and functional status in terminal-stage cancer patients receiving palliative care. Participants are divided into two groups: the intervention group receives supervised breathing exercises by a physiotherapist, while the control group is given an informational brochure without any physical guidance.

The primary objective is to determine whether supervised breathing exercises provide significant improvements in symptom control and functionality compared to usual care. Assessments are made before and after the intervention using validated tools including the Edmonton Symptom Assessment System (ESAS-r), the Cancer Dyspnea Scale (CDS), and the Visual Analog Scale (VAS) for pain.

The study aims to contribute to the clinical evidence supporting non-pharmacological interventions in palliative care and to offer practical approaches for improving quality of life in terminally ill cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving palliative care, who are part of this treatment process and considered eligible for the study.
* Patients diagnosed with Stage 4 cancer, included in the study due to their advanced cancer stage.
* Patients with oxygen saturation levels below 95% in room air, who are deemed appropriate for monitoring respiratory function due to this condition.
* Participants must be able to effectively communicate during the study period.
* Individuals who agree to participate in the study must provide written or verbal consent, which is a mandatory criterion for ethical compliance.

Exclusion Criteria:

* Patients who are unconscious and unable to participate in the study. Individuals under the age of 18.
* Patients dependent on a ventilator.
* Patients with serious health issues, such as uncontrolled hypertension and dyspnea.
* Patients with other significant health problems that prevent participation in the research program.
* Patients with medical conditions requiring drainage treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
dyspnea | From enrollment to the end of treatment at 1 weeks
  Dyspnea severity will be assessed using the Edmonton Symptom Assessment System - revised (ESAS-r) dyspnea item. This is a numeric rating scale ranging from 0 to 10, where 0 indicates no shortness of breath and 10 indicates the worst possible shortness of breath. The outcome will evaluate changes in dyspnea severity following a structured breathing exercise intervention.
Functionality | From enrollment to the end of treatment at 1 weeks
  Functionality will be measured using the Edmonton Symptom Assessment System - revised (ESAS-r) physical well-being domain. The ESAS-r is a validated self-report instrument in which patients rate symptom severity on a scale from 0 to 10, with 0 indicating no impairment and 10 indicating the worst possible level of functional impairment. This outcome assesses changes in participants' ability to perform daily activities such as walking, dressing, and self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Yaşar Gül BALTACI, Prof. Dr., Study Director — İstanbul Atlas University, Department of Physical Medicine and Rehabilitation
Locations (1):
- Eyupsultan State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
This clinical trial evaluates the effects of structured respiratory exercises on pain, dyspnea, and physical functionality in terminal-stage cancer patients under palliative care. It is a single-arm interventional study with pre- and post-intervention assessments. Participants perform pursed-lip and diaphragmatic breathing exercises under physiotherapist supervision for one week. The primary outcomes are changes in pain and dyspnea, measured using ESAS-r and CDS. Secondary outcomes include functional status assessed via standardized tools. Data are collected at baseline and after the intervention. The study follows the Declaration of Helsinki and has received institutional ethical approval. Results aim to support the use of non-pharmacological methods in enhancing the quality of life for patients in end-of-life care.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The intervention will be applied for 1 week per participant. Respiratory exercises will be conducted daily for 5 consecutive days. Baseline and post-intervention assessments will be performed at the beginning and end of the week, respectively.
Access Criteria: De-identified individual participant data (IPD) may be made available upon reasonable request for academic or research purposes. Access requires submission of a detailed proposal and prior approval by the study investigator. Requests can be sent to yildiz.fatmanur@hotmail.com.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT07164352/Prot_SAP_000.pdf
  • Informed Consent Form (2025-08-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT07164352/ICF_001.pdf